CLINICAL TRIAL: NCT01191762
Title: The Effect of Sevelamer Carbonate on Critical Variables in the Pathogenesis of Secondary Hyperparathyroidism
Brief Title: Sevelamer and Secondary Hyperparathyroidism in Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kenneth R. Phelps, M.D. (Individual)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Kenneth R. Phelps, M.D., Principal Investigator, Phelps, Kenneth R., M.D.
Organization: Phelps, Kenneth R., M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhelpsK
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Hyperparathyroidism; Chronic Kidney Disease
Keywords: secondary hyperparathyroidism; phosphate; calcium; chronic kidney disease
MeSH Terms: conditions — Hyperparathyroidism; Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevelamer carbonate (Active Comparator): 2400 mg (3 pills) with each meal
  Interventions: Drug: sevelamer carbonate
- placebo control (Placebo Comparator): 3 placebo tablets with each meal; tablets are identical to sevelamer carbonate 800 mg tablets.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sevelamer carbonate — 2400 mg with each meal for 4 weeks
  Other Names: Renvela (Genzyme)
  Arms: sevelamer carbonate
Drug: placebo — 3 tablets with each meal
  Arms: placebo control

SUMMARY:
The hypothesis underlying this study is that phosphate interferes with PTH-mediated calcium reabsorption in the distal nephron and thereby necessitates supranormal [PTH]to maintain normocalcemia in chronic kidney disease. This study will examine the hypothesis with measures of phosphate homeostasis and calcium reabsorption. A double-blind trial of the intestinal phosphate binder sevelamer carbonate will be employed to examine whether reductions in phosphate influx alter distal nephron phosphate concentration and the [PTH] required for calcium reabsorption in the expected manner.

DETAILED DESCRIPTION:
The parathyroid hormone concentration ([PTH)] rises as glomerular filtration rate (GFR) falls. This almost universal phenomenon is called secondary hyperparathyroidism (SHPT). [PTH] rises with dietary phosphate in chronic kidney disease. [PTH] also rises with stable dietary phosphate as GFR falls. The mechanism underlying these phenomena is unknown.

We hypothesize that phosphate exerts its effect on [PTH] in the cortical distal nephron (CDN). Ordinarily, intestinal phosphate absorption does not fall in proportion to GFR as chronic kidney disease (CKD) progresses. Consequently, the concentration of phosphate increases in the cortical distal nephron (CDN), where PTH regulates tubular calcium reabsorption. We speculate that increased [P]cdn reduces the concentration of free calcium through complexation, and thereby necessitates high [PTH] for achievement of calcium reabsorption sufficient to maintain normocalcemia. We can show algebraically that [P]cdn is proportional to the ratio EP/Ccr, where EP is the urinary excretion rate of phosphate and Ccr is creatinine clearance, a surrogate for GFR. EP/Ccr can be calculated from measurements in aliquots of serum and urine as [P]u[cr]s/[cr]u. If our hypothesis is correct, we anticipate that [PTH] will be proportional to EP/Ccr in CKD, and that delta [PTH] will be proportional to delta EP/Ccr obtained with sequential determinations.

We will study 30 patients with CKD and a comparable number of controls. All subjects will have normocalcemia. Controls will be seen once for informed consent, and once in the fasting state between 8:00 a.m. and 10:00 a.m. for collection of urine and blood specimens.

Patients with CKD will be seen at five visits at intervals of four weeks. At the first visit, we will obtain informed consent and obtain a specimen for measurement of 25-hydroxyvitamin D (25OHD). At visits 2-5, we will obtain necessary specimens to measure concentrations of PTH, fibroblast growth factor 23 (FGF23), 25OHD, and 1,25-dihyroxyvitamin D (1,25(OH)2D). We will also measure ionized and ultrafilterable calcium, creatinine, and phosphorus in serum and calcium, phosphorus, and creatinine in urine. These measurements will enable us to follow the effects of interventions on hormone concentrations and parameters of calcium and phosphorus homeostasis.

At visit 2 we will prescribe vitamin D in accordance with [25OHD] obtained at visit 1. For [25OHD] < 32 ng/mL, doses will be 50,000 units/d of D2 for one week, followed by 2000 mg/d of D2 for 3 weeks. For [25OHD] > 32 ng/mL, the dose will be D3 2000 mg/d for four weeks. The purpose of this intervention is to minimize the likelihood that vitamin D insufficiency or deficiency contributes to SHPT.

At visit 3, we will instruct patients in a phosphate-restricted diet. At visit 4 we will quantify the metabolic effects of the diet, and will randomly assign patients to receive either placebo or sevelamer carbonate 800 mg tablets, 3 with each meal. At visit 5, we will quantify the effects of the two interventions on parameters of calcium and phosphate homeostasis and on hormone concentrations. We will view positive regressions of [PTH] on EP/Ccr and of ∆[PTH] on ∆EP/Ccr as evidence for our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* eGFR < 60 ml/min
* age at least 18 years

Exclusion Criteria:

* any primary parathyroid disease

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R. Phelps, M.D., Principal Investigator — Stratton VAMC, Albany, NY
Locations (1):
- Stratton Veterans Affairs Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Phelps KR, Mason DL. Parathyroid Hormone, Fibroblast Growth Factor 23, and Parameters of Phosphate Reabsorption. Am J Nephrol. 2018;47(5):343-351. doi: 10.1159/000489270. Epub 2018 May 18. PMID 29779023
- [Derived] Phelps KR, Mason DL, Stote KS. Phosphate homeostasis, parathyroid hormone, and fibroblast growth factor 23 in stages 3 and 4 chronic kidney disease. Clin Nephrol. 2016 May;85(5):251-61. doi: 10.5414/CN108686. PMID 26951967
- [Derived] Phelps KR, Mason DL. Parameters of phosphorus homeostasis at normal and reduced GFR: theoretical considerations. Clin Nephrol. 2015 Mar;83(3):167-76. doi: 10.5414/cn108367. PMID 25685872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with eGFR < 60 were recruited from renal clinics and randomized to receive 3 tablets of sevelamer or placebo with each meal for four weeks.
Pre-assignment Details: Randomization was preceded by a 4-week course of vitamin D (dose determined by plasma [25OHD]) and then by a 4-week period of dietary phosphate restriction. The phosphate restriction was continued through the therapeutic trial.
Groups:
- Sevelamer Carbonate: 2400 mg (3 pills) with each meal
  sevelamer carbonate : 2400 mg with each meal for 4 weeks
- Placebo Control: 3 placebo tablets with each meal; tablets are identical to sevelamer carbonate 800 mg tablets.
  placebo : 3 tablets with each meal
Period: Overall Study
Arm/Group | Sevelamer Carbonate | Placebo Control
Started | 15 | 15
Completed | 14 (One subject dropped out on the 3rd treatment day because of gastrointestinal complaints.) | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Post-treatment data were not obtained from patient who withdrew on third treatment day.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevelamer Carbonate | Placebo Control | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (8.5) | 70.1 (10.5) | 71.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Fractional Change in [PTH] in CKD After a 4-week Course of Sevelamer Carbonate
Description: This outcome measure documented the effect of intestinal phosphate-binding on [PTH]. Fractional change was calculated as ([PTH]post - [PTH]pre)/[PTH]pre, where 'pre' and 'post' referred respectively to baseline [PTH] (before treatment) and [PTH] after four weeks of treatment. Reductions were cited as negative numbers, and increments were cited as positive numbers.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: percentage of baseline [PTH]
Arm/Group | Sevelamer Carbonate | Placebo Control
Number analyzed (Participants) | 14 | 15
percentage of baseline [PTH] | -11.7 (5.8) | 16.4 (10.0)

ADVERSE EVENTS:
Arm/Group | Sevelamer Carbonate | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevelamer Carbonate (N=15) | Placebo Control (N=15)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — The patient complained of nausea and upset stomach from the inception of his treatment.

LIMITATIONS AND CAVEATS:
All intended measurements were made. The desired number of participants was recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No